CLINICAL TRIAL: NCT05028634
Title: A Phase 3b, Multicenter, Open-label Study to Evaluate the Immune Response to, and the Safety of, Vaccines in Participants With Relapsing Forms of Multiple Sclerosis Who Receive Oral Ozanimod Compared to Non-pegylated Interferon (IFN)-β or No Disease Modifying Therapy
Brief Title: Safety Study to Evaluate Immune Response of Vaccines in Participants With Relapsing Forms of Multiple Sclerosis Who Receive Ozanimod Compared to Non-Pegylated Interferon (IFN)-β or No Disease Modifying Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPC-1063-MS-010; 2021-001847-28 (EudraCT Number)
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Ozanimod; Relapsing-remitting multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - Ozanimod (Experimental): Comprises of participants received oral ozanimod will be administered tetanus, diphtheria, and acellular pertussis vaccine (Tdap), pneumococcal polysaccharide vaccine (PPSV23), and the seasonal inactivated influenza vaccine
  -Enrollment is closed for this cohort
  Interventions: Biological: Tetanus, diphtheria, and acellular pertussis vaccine; Biological: Pneumococcal polysaccharide vaccine; Biological: Seasonal influenza vaccine
- Cohort 1 - non-pegylated interferon-β or no disease modifying therapy (Experimental): Comprises of participants received either non-pegylated interferon-β (IFN-β) or no disease modifying therapy (DMT) will be administered tetanus, diphtheria, and acellular pertussis vaccine (Tdap), Pneumococcal polysaccharide vaccine (PPSV23), and the seasonal inactivated influenza vaccine
  -Enrollment is closed for this cohort
  Interventions: Biological: Tetanus, diphtheria, and acellular pertussis vaccine; Biological: Pneumococcal polysaccharide vaccine; Biological: Seasonal influenza vaccine
- Cohort 2 - Ozanimod (Experimental): Comprises of participants received oral ozanimod will be administered tetanus, diphtheria, and acellular pertussis vaccine (Tdap), and pneumococcal polysaccharide vaccine (PPSV23).
  Interventions: Biological: Tetanus, diphtheria, and acellular pertussis vaccine; Biological: Pneumococcal polysaccharide vaccine
- Cohort 2 - non-pegylated interferon-β or no disease modifying therapy (Experimental): Comprises of participants received either non-pegylated interferon-β (IFN-β) or no disease modifying therapy (DMT) will be administered tetanus, diphtheria, and acellular pertussis vaccine (Tdap) and Pneumococcal polysaccharide vaccine (PPSV23).
  Interventions: Biological: Tetanus, diphtheria, and acellular pertussis vaccine; Biological: Pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: Tetanus, diphtheria, and acellular pertussis vaccine — Tdap
  Other Names: Tdap
Biological: Pneumococcal polysaccharide vaccine — PPSV23
  Other Names: PPSV23
Biological: Seasonal influenza vaccine — Seasonal influenza vaccine
  Arms: Cohort 1 - Ozanimod; Cohort 1 - non-pegylated interferon-β or no disease modifying therapy

SUMMARY:
This study is designed to provide data on the immune response and safety of administering vaccines to relapsing multiple sclerosis (RMS) participants taking ozanimod compared to controls taking interferon-beta's or receiving no disease modifying therapies (DMTs). The data of this study will support the labels for ozanimod in multiple sclerosis (MS) because the effect of ozanimod on the vaccination response of MS participants is of interest to participants and prescribers.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of multiple sclerosis (MS) according to the 2017 revision of the McDonald diagnostic criteria and has relapsing forms of multiple sclerosis (RMS): relapsing-remitting MS (RRMS) or secondary progressive MS with active disease based on recent clinical relapse or MRI lesion activity.

Exclusion Criteria:

* Participant has history of cancer, including solid tumors and hematological except for basal cell cancer of the skin and carcinoma in situ of the cervix, which are exclusionary if they have not been excised and resolved.
* Participant has a history of or currently active primary or secondary immunodeficiency.
* Participant has severely compromised cardiac or pulmonary function for which a systemic hypersensitivity reaction to any of the vaccines would pose a significant risk.
* Participant has received the seasonal influenza vaccine for the 2021/2022 influenza season prior to Day 1, or history of influenza vaccine for the 2020/2021 influenza season within 6 months prior to Day 1.
* Participant has previous treatment with one of the following medications or interventions within the corresponding timeframe described as follows:

  * Any systemic immunosuppressive treatments with potential overlapping effects with the baseline of this study. Corticosteroids that are by non-systemic routes (e.g., topical, inhaled, intra-articular) are allowed.
* History of treatment with IV immunoglobulin (IVIg) or plasmapheresis within 4 weeks prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (29):
  - Stanford University, Palo Alto, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Hartford Healthcare CT, Southington, Connecticut
  - University of Florida Health, Gainesville, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Accel Research Sites - Brain and Spine Institute of Port Orange - ERN - PPDS, Port Orange, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Consultants In Neurology, Northbrook, Illinois
  - Local Institution - 111, Kansas City, Kansas
  - CPFCC Neurology Research Dept., Overland Park, Kansas
  - Neuromedical Clinic of Central LA, Alexandria, Louisiana
  - Neurology Center of New England P.C., Foxborough, Massachusetts
  - Michigan State University MS Clinic, East Lansing, Michigan
  - Shapiro Center for MS at the Minneapolis Clinic of Neurology, Minneapolis, Minnesota
  - Neurology Associates PC, Lincoln, Nebraska
  - Jersey Shore MS Center, Neptune City, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - South Shore Neurology Associates, Inc, Patchogue, New York
  - Asheville Neurology Specialists PA, Asheville, North Carolina
  - Lake Norman Neurology, Mooresville, North Carolina
  - Local Institution - 105, Canton, Ohio
  - Velocity Clinical Research - Cleveland - ERN - PPDS, Cleveland, Ohio
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - Hope Neurology MS Center, Knoxville, Tennessee
  - Central Texas Neurology Consultants PA, Round Rock, Texas
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - Vaught Neurological Services, PLLC, Crab Orchard, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (4):
  - Local Institution - 200, Bochum
  - Local Institution - 201, Dresden
  - Local Institution - 206, Mannheim
  - Local Institution - 204, Rostock

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As pre-specified per protocol, Cohort 1 and Cohort 2 are pooled per the following treatment groups.
  i. Ozanimod treatment group ii. Non-Ozanimod treatment group
Groups:
- Ozanimod: Participants with relapsing forms of Multiple Sclerosis (MS) who received Oral Ozanimod were administered with regimen of Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis, Adsorbed (Tdap) vaccine, Pneumococcal polysaccharide (PPSV23), and the seasonal inactivated influenza vaccine on Day 1.
- Non-Ozanimod: Participants with relapsing forms of Multiple Sclerosis (MS) who have received either non-pegylated interferon-β (IFN-β) or no disease modifying therapy (DMT) and already received the seasonal inactivated influenza vaccine receive regimen of Tdap and PPSV23 vaccine only on Day 1.
Period: Overall Study
Arm/Group | Ozanimod | Non-Ozanimod
Started | 30 | 33
Completed | 30 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozanimod | Non-Ozanimod | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (9.03) | 46.8 (6.83) | 45.0 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 24 | 29 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Immune Serological Response Criteria to Tetanus Toxoid Antigen
Description: Serologic response to tetanus toxoid criteria are as follows - if pre vaccination antibody titer is ≤0.10 IU/mL, post-vaccination level ≥0.40 IU/mL; if pre-vaccination antibody titer is >0.10 IU/mL and ≤2.7 IU/mL, at least a 4-fold increase in titer; if pre-vaccination antibody titer is>2.7 IU/mL, at least a 2-fold increase in titer.
Time Frame: Day 28
Population: Modified Intent-to-Treat (mITT) Population consists of all participants who received at least one vaccination and summarized according to their initial treatment status (ozanimod vs. non-ozanimod) regardless of systemic use of corticosteroids. Participants with data available at the specified timepoint are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 32
percentage of participants | 10 | 53.1

2. Primary Outcome: Percentage of Participants Meeting Immune Serological Protection Criteria to Tetanus Toxoid Antigen
Description: Participants with Serological protection to tetanus toxoid have anti-tetanus toxoid IgG concentration >= 0.1 International Units per milliliter (IU/mL).
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 33
percentage of participants | 100 | 100

3. Secondary Outcome: Percentage of Participants With Serologic Response to Pneumococcal Polysaccharide Vaccine (PPSV23)
Description: Serological response to PPSV23 was defined as the percentage of participants with a ≥2-fold increase in anti-pneumococcal polysaccharide vaccine titer in >5 of the indicated serotypes - 3, 6B, 9N, 11A, 14, 19A, 19F, 22F and 23F
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 29 | 32
percentage of participants | 69.0 | 87.5

4. Secondary Outcome: Percentage of Participants With Serologic Protection Against Pneumococcal Polysaccharide Vaccine (PPSV23)
Description: Serological protection against PPSV23 was defined as the percentage of participants with Anti-pneumococcal polysaccharide IgG concentration >= 1.3 μg/mL in the indicated serotypes - 3, 6B, 9N, 11A, 14, 19A, 19F, 22F and 23F associated with increased risk of invasive and/or severe disease, including death.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 32
percentage of participants | 66.7 | 71.9

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events include events with onset date on or after the study medication first dose date until end of study visit after the vaccine administration. Serious AEs was defined as is any AE occurring at any dose of vaccination from Day 1 to the end of the study that results in death, Is life-threatening (ie, in the opinion of the Investigator, the subject is at immediate risk of death from the AE), Requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or constitutes an important medical event.
Time Frame: Day 1 to Day 28
Population: Modified Intent-to-Treat (mITT) Population consists of all participants who received at least one vaccination and summarized according to their initial treatment status (ozanimod vs. non-ozanimod) regardless of systemic use of corticosteroids.
Measure: Count of Participants; unit: Participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 33
Participants
  AEs | 11 | 11
  SAEs | 0 | 0
  Moderate or Severe AEs | 2 | 4
  AEs leading to Death | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormalities in Blood Chemistry Parameters
Description: Blood samples were collected to assess laboratory parameters
Time Frame: Day 1 to Day 28
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 33
Participants
  Alanine Transaminase (ALT) OR Aspartate aminotransferase (AST) > 1X Upper Limit of Normal (ULN) | 6 | 7
  ALT or AST > 2XULN | 1 | 1
  ALT OR AST > 3XULN | 0 | 0
  ALT OR AST > 5XULN | 0 | 0
  ALT OR AST > 10XULN | 0 | 0
  Gamma-glutamyl transferase (GGT) OR Alkaline Phosphatase (ALP) > 1XULN | 7 | 4
  GGT OR ALP > 2.5XULN | 2 | 0
  GGT OR ALP > 5XULN | 1 | 0
  GGT OR ALP > 20XULN | 0 | 0
  TOTAL BILIRUBIN > 1XULN | 0 | 1
  TOTAL BILIRUBIN > 1.5XULN | 0 | 1
  TOTAL BILIRUBIN > 2XULN | 0 | 0
  TOTAL BILIRUBIN > 3XULN | 0 | 0
  TOTAL BILIRUBIN > 10XULN | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormalities in Blood Hematology Parameters
Description: Blood samples were collected to assess laboratory parameters
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 29 | 33
Participants
  ABSOLUTE LYMPHOCYTE COUNT (ALC) < 0.2 (x10E9/L) | 1 | 0
  ABSOLUTE NEUTROPHIL COUNT (ANC) < 0.5 (x10E9/L) | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT (ANC) < 1 (x10E9/L) | 0 | 0
  TOTAL WBC > 20 (x10E9/L) | 0 | 0

8. Secondary Outcome: Change From Baseline in Blood Chemistry Parameters - Sodium; Potassium; Chloride; Calcium; Magnesium; Phosphate; Blood Urea Nitrogen; Glucose
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 31
mmol/L
  Sodium | -0.7 (1.90) | -0.3 (2.56)
  Potassium | -0.14 (0.637) | -0.08 (0.315)
  Chloride: number analyzed (Participants) | 28 | 31
  Chloride | -0.9 (5.19) | 0.2 (2.63)
  Calcium: number analyzed (Participants) | 28 | 31
  Calcium | -0.044 (0.0881) | -0.015 (0.0888)
  Magnesium: number analyzed (Participants) | 28 | 31
  Magnesium | -0.003 (0.0572) | -0.001 (0.0549)
  Phosphate: number analyzed (Participants) | 28 | 31
  Phosphate | -0.011 (0.2197) | -0.041 (0.1640)
  Blood Urea Nitrogen: number analyzed (Participants) | 28 | 31
  Blood Urea Nitrogen | 0.044 (1.1424) | 0.165 (1.1542)
  Glucose: number analyzed (Participants) | 28 | 31
  Glucose | 0.28 (0.845) | 0.08 (0.946)

9. Secondary Outcome: Change From Baseline in Blood Chemistry Parameters - Creatinine; Bilirubin; Direct Bilirubin
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 31
umol/L
  Creatinine: number analyzed (Participants) | 28 | 31
  Creatinine | -1.1 (9.64) | -0.6 (9.77)
  Bilirubin: number analyzed (Participants) | 27 | 31
  Bilirubin | 0.4 (2.81) | 0.1 (3.09)
  Direct Bilirubin: number analyzed (Participants) | 26 | 30
  Direct Bilirubin | 0.0 (0.20) | 0.0 (0.18)

10. Secondary Outcome: Change From Baseline in Blood Chemistry Parameters - Albumin
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 30 | 31
g/L | -0.2 (2.67) | -0.8 (2.91)

11. Secondary Outcome: Change From Baseline in Blood Chemistry Parameters - Alkaline Phosphatase
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 28 | 31
IU/L | 2.9 (14.48) | -1.1 (8.73)

12. Secondary Outcome: Change From Baseline in Blood Chemistry Parameters - Alanine Aminotransferase; Aspartate Aminotransferase; Gamma Glutamyl Transferase
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 28 | 33
U/L
  Alanine Aminotransferase: number analyzed (Participants) | 28 | 31
  Alanine Aminotransferase | 3.5 (8.88) | 1.4 (5.08)
  Aspartate Aminotransferase: number analyzed (Participants) | 25 | 31
  Aspartate Aminotransferase | 2.1 (3.77) | 0.9 (5.64)
  Gamma Glutamyl Transferase: number analyzed (Participants) | 28 | 31
  Gamma Glutamyl Transferase | 3.2 (23.09) | 0.6 (8.39)

13. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Erythrocytes
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 24 | 31
10^12 cells per liter | -0.06 (0.191) | -0.07 (0.265)

14. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Leukocytes; Basophils; Eosinophils; Lymphocytes; Monocytes; Neutrophils; Platelets
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 24 | 31
10^9 cells per liter
  Leukocytes: number analyzed (Participants) | 23 | 31
  Leukocytes | 0.58 (1.271) | 0.33 (1.298)
  Basophils: number analyzed (Participants) | 21 | 31
  Basophils | -0.013 (0.0320) | -0.007 (0.0253)
  Eosinophils: number analyzed (Participants) | 21 | 31
  Eosinophils | 0.038 (0.2872) | 0.013 (0.1531)
  Lymphocytes: number analyzed (Participants) | 21 | 31
  Lymphocytes | 0.046 (0.1806) | 0.021 (0.3580)
  Monocytes: number analyzed (Participants) | 21 | 31
  Monocytes | -0.021 (0.1734) | 0.025 (0.1506)
  Neutrophils: number analyzed (Participants) | 21 | 31
  Neutrophils | 0.480 (1.1208) | 0.218 (1.2622)
  Platelets: number analyzed (Participants) | 24 | 28
  Platelets | -5.3 (37.08) | 1.4 (36.33)

15. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Basophils/Leukocytes; Eosinophils/Leukocytes; Lymphocytes/Leukocytes; Monocytes/Leukocytes; Neutrophils/Leukocytes
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 21 | 31
percentage
  Basophils/Leukocytes | -0.34 (0.528) | -0.14 (0.442)
  Eosinophils/Leukocytes | 0.05 (3.919) | 0.05 (1.950)
  Lymphocytes/Leukocytes | 0.17 (3.675) | -1.35 (6.883)
  Monocytes/Leukocytes | -0.97 (3.135) | 0.03 (2.192)
  Neutrophils/Leukocytes | 1.09 (6.750) | 1.40 (7.177)

16. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Hemoglobin; Erythrocytes Mean Corpuscular HGB Concentration
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 24 | 31
g/L
  Hemoglobin | -1.9 (5.67) | -2.9 (7.14)
  Erythrocytes Mean Corpuscular HGB Concentration: number analyzed (Participants) | 23 | 31
  Erythrocytes Mean Corpuscular HGB Concentration | 1.2 (9.81) | 0.2 (9.16)

17. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 23 | 31
fL | -0.3 (2.25) | -0.5 (1.95)

18. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to assess laboratory parameters.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 24 | 31
pg/cell | -0.1 (0.65) | -0.1 (0.72)

19. Secondary Outcome: Change From Baseline in Blood Hematology Parameters - Hematocrit
Description: Blood samples were collected to assess laboratory parameters. Participants with baseline and post-baseline data available at the specified timepoint are included in the analysis.
Time Frame: Baseline (Day 1) and End of Study (Day 28)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Ozanimod | Non-Ozanimod
Number analyzed (Participants) | 23 | 31
Proportion of red blood cells in blood | -0.007 (0.0226) | -0.010 (0.0270)

ADVERSE EVENTS:
Time Frame: All cause mortality and Non Serious and Serious adverse events were collected from first dose (Day 1) until end of study visit (Day 28).
Description: As pre-specified per protocol, Cohort 1 and Cohort 2 are pooled per the following treatment groups.
  i. Ozanimod treatment group ii. Non-Ozanimod treatment group Modified Intent-to-Treat (mITT) Population consists of all participants who received at least one vaccination and summarized according to their initial treatment status (ozanimod vs. non-ozanimod) regardless of systemic use of corticosteroids.
Arm/Group | Ozanimod | Non-Ozanimod
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 5/30 | 7/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod (N=30) | Non-Ozanimod (N=33)
Fatigue (General disorders) | 2 | 1
Injection site pain (General disorders) | 1 | 4
COVID-19 (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT05028634/Prot_SAP_000.pdf